CLINICAL TRIAL: NCT00603616
Title: A Randomized, Prospective, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Safety and Efficacy of Rifaximin for the Treatment of Moderate to Severe Crohn's Disease
Brief Title: Induction of Clinical Response Using Rifaximin in Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scott Lee (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Scott Lee, Professor, University of Washington
Organization: University of Washington (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 32871; 32871 (Other: University of Washington)
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Crohn's Disease
Keywords: Inflammatory Bowel Disease; Crohn disease; Crohn's disease; Rifaximin
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- 1 (Placebo Comparator): Placebo pills
  Interventions: Drug: Placebo Comparator
- 2 (Active Comparator): Rifaximin
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Placebo Comparator — Matching oral placebo pills to be taken twice daily for a total of 8 weeks
  Arms: 1
Drug: Rifaximin — Oral rifaximin 550mg to be taken twice daily for a total of 8 weeks
  Other Names: Xifaxan
  Arms: 2

SUMMARY:
Antibiotics have been used to treat Crohn's disease symptoms with the best studied antibiotics being Cipro and Flagyl. Rifaximin is a poorly absorbed oral antibiotic that is FDA approved for travelers' diarrhea. It works by inhibiting bacterial reproduction. It is very poorly absorbed and over 97% of the drug taken orally is excreted in the feces.

The purpose of this study is to evaluate the potential benefits and safety of Rifaximin for the treatment of moderate to severe symptoms of Crohn's Disease.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a debilitating chronic inflammatory disease conventionally categorized into Crohn's disease (CD) and Ulcerative Colitis (UC). CD affects nearly 630,000 people in North America with up to 50,000 new people being diagnosed every year. It is a chronic debilitating disease characterized by abdominal pain, malnutrition, bloody diarrhea, fistula formation, intestinal perforations and strictures, and even extra-intestinal manifestations such as joint pains and skin rashes. Nearly 80% of people with CD will need surgical treatment at some point in their disease process. The majority of CD subjects are diagnosed in young adulthood thereby subjecting them to many decades of discomfort and medical intervention.

Antibiotics have been used to treat CD with variable response rates. The basis for antibiotic therapy is that breakdown of the integrity of the mucosal barrier in the gastrointestinal (GI) tract leads to a heightened inflammatory response to commensurate luminal bacteria. By changing the composition or bacterial load in the intestinal lumen, it may be possible to alter the immune response. Ciprofloxacin (Cipro) and metronidazole (Flagyl) are the best studied antibiotics that have shown efficacy, but the effect is temporal and long term use can lead to serious side effects. Rifaximin is a recent FDA approved antibiotic with broad spectrum of activity, excellent safety profile, and minimal absorption from the GI tract. Open label and small studies in IBD subjects show response rates up to 80% in CD subjects. These studies were limited however in that they were not randomized placebo controlled trials.

The investigators propose to conduct a randomized placebo controlled crossover trial of rifaximin in CD subjects to assess initial clinical response compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 80 years of age, inclusive, that can themselves provide written, informed consent and authorization of use of protected health information prior to any study-related procedures and who are, in the opinion of the investigator(s), likely to comply with all the requirements of the study
* Subjects must have a prior diagnosis of CD established by endoscopy and clinical parameters as determined by the investigator(s) for at least 3 months prior to randomization
* Subjects must be able to participate in all required follow-up visits and fill out all related documentation (e.g. symptom diary)
* Subjects currently with moderately active disease defined as a CDAI 250-450
* Concomitant medications:

  * If subjects are taking sulfasalazine or 5-ASA products prior to entry, the dose must be stable for at least 4 weeks prior to the randomization
  * If subjects are on azathioprine, 6-mercaptopurine, or methotrexate, they will have had to be on a stable dosage for at least 8 weeks
  * Subjects are allowed to be on corticosteroids at a dose equivalent to 20 mg or less of prednisone, IF the dose has been stable for a minimum of 2 weeks. Steroids must be held stable throughout the induction portion of the study. The maximum dose of budesonide must not exceed 9mg per day and must also have been stable for a minimum of 2 weeks.
  * No oral or intravenous antibiotics within 4 weeks prior to randomization
  * No current or past use of biological treatment within 6 weeks of randomization into study (e.g. infliximab)
  * If subjects have previously been on any of the above products but are no longer taking them, they should not have received any of the relevant therapeutic products within 4 weeks prior to randomization
  * No other experimental or non-FDA approved medications are allowed. If the subject has previously been on an experimental therapy, they must have not received the therapy within the prior 8 weeks prior to randomization
  * Subjects on concomitant medications for CD will not be allowed to change dosages during the study
* If subjects are at increased risk of colorectal cancer (defined as having an 8-year history of pan-colitis or 12 year history of left sided colitis), they will need to have undergone a colonoscopy with pan-colonic surveillance biopsies within 2 years of the screening visit. The biopsies must be negative for dysplasia
* Female or male subjects who are surgically sterilized or who are prepared to and agree to practice a double-barrier form of birth control from the screening visit through 30 days (females) and 30 days (males), respectively, from the last dose of study medication. Females who are more than 12 months post-menopausal are also eligible to participate in the study

Exclusion Criteria:

* Evidence of active infection which may include any of the following

  * Febrile ( > 38.5ºC)
  * Positive blood culture within 2 weeks prior to randomization
  * Evidence of toxic megacolon or abscess
  * Positive stool culture for enteric pathogens, pathogenic ova or parasite, or a positive assay for C. difficile toxin at screening
* Subjects with CDAI > 450
* Any current use or use within the last 8 weeks of an investigational drug
* Current or past use (within past 12 wks) of biological treatment
* Current or use within the last 4 weeks of any oral or intravenous antibiotic
* Anticipated increased dosage of any medication to treat CD
* Anticipated need for surgery within 12 weeks
* Known obstructive diseases of the gastrointestinal system
* Medical conditions requiring in-patient hospitalization
* Proctocolectomy, total colectomy, ileostomy, or stoma
* Severe cardiopulmonary disease:

  * Congestive heart failure (NYHA Class III or IV)
  * Severe cardiovascular or peripheral vascular disease
  * Myocardial infarction, percutaneous coronary intervention, or bypass surgery within the past 6 months
* Significant liver disease:

  * Levels of SGOT [AST], SGPT [ALT], or alkaline phosphatase > 2.5x the upper limit of the normal range for the laboratory performing test
  * History of cirrhosis
* Renal insufficiency, defined as serum creatinine > 150% of the upper limit of the normal range for the laboratory performing the test
* Abnormal hematology parameters defined as severe anemia with hemoglobin < 8.5 g/dL and/or white blood cell count of < 3,500/ul
* Malignancy within the past 2 years other than surgically cured skin carcinoma or cervical dysplasia (CIN I-II)
* History of dysplasia or carcinoma of the colon
* Pregnant, lactating, or planning to become pregnant during the course of the investigational study
* Known history of allergic reaction to rifaximin or allergy to any of the rifamycin antimicrobial agents (which include rifampin, rifabutin, and rifapentine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-11; Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of rifaximin 550 mg bid compared to placebo in achieving clinical response in moderate to severe Crohn's Disease (CD) subjects as determined by a > 100 point decrease in the Crohn's Disease Activity Index (CDAI) | 8 weeks

SECONDARY OUTCOMES:
Evaluate the efficacy of rifaximin compared to placebo at inducing clinical remission in CD subjects | 8 weeks
Evaluate the safety profile of rifaximin in subjects with active CD | 16 weeks for those subjects who do not cross over, 32 weeks for those who do cross over
Evaluate the effect rifaximin has on the quality of life in subjects with CD compared to placebo | 8 weeks
Evaluate if there are any clinical parameters which might predict response to rifaximin | 8 weeks
Compare mean changes in CDAI scores between rifaximin and placebo treated subjects | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Lee, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No